CLINICAL TRIAL: NCT00600353
Title: Combined Use of Multi-Day Doses of Palonosetron and Aprepitant With Low Doses Dexamethasone in Prevention of Nausea and Emesis Among Patients With Multiple Myeloma and Lymphoma Undergoing Autologous Stem Cell Transplant: A Pilot Study
Brief Title: Multi-day Doses in Prevention of Nausea and Emesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10862; NCT00631930 (obsolete NCT alias)
Record Dates: First submitted 2008-01-07; First posted 2008-01-25 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Myeloma, Plasma-Cell; Lymphoma, Malignant
Keywords: nausea; cancer; CINV
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Nausea; Neoplasms | interventions — Palonosetron; Aprepitant; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melphalan, dexamethasone, aprepitant, palonosetron (Experimental): Group A: Subjects with Multiple Myeloma
  * Conditioning regimen, over a 7 day period, includes:
  * Melphalan 70-100 mg, Dexamethasone 4 mg IV push, Aprepitant 125 mg PO, Palonosetron 0.25 mg IV over 30 seconds, Aprepitant 80 mg PO, Dexamethasone 4 mg IV and Lorazepam 1 mg IV x 1 dose 30 minutes prior to stem cell infusion
  Group B: Subjects with Lymphoma
  * Conditioning regimen, over a 7 day period, includes: (BEAC)
  * BCNU 300 mg/m2 IV x 1,Cytarabine 100 mg/m2 IV BID, Etoposide 100 mg/m2 IV BID, administer after, Cyclophosphamide 35 mg/kg QD, Dexamethasone 4 mg IV push, Aprepitant 125 mg PO, Palonosetron 0.25 mg IV over 30 seconds, Aprepitant 80 mg PO, Lorazepam 1 mg IV x 1 dose 30 minutes prior to stem cell transplant
  Interventions: Drug: Palonosetron; Drug: Aprepitant; Drug: Dexamethasone

INTERVENTIONS:
Drug: Palonosetron — Palonosetron 0.25 mg IV over 30 seconds
  Other Names: Aloxi
Drug: Aprepitant — Aprepitant 125 mg PO and Aprepitant 80 mg PO
  Other Names: Emend
Drug: Dexamethasone — Dexamethasone 4 mg IV and Dexamethasone 4 mg IV push
  Other Names: Decadron

SUMMARY:
To assess emetic responses to multi-day doses of Palonosetron and Aprepitant and low dose dexamethasone +/- Prochlorperazine among patients with multiple myeloma and lymphoma undergoing autologous HSCT utilizing the Multinational Association for Supportive Care in Cancer (MASCC) Antiemesis Tool (MAT).

DETAILED DESCRIPTION:
The use of high doses of chemotherapy and autologous stem cell transplant has been shown to prolong disease control among patients with multiple myeloma and patients with lymphomas that have relapsed or recurred. Patients who receive autologous stem cell transplants have their own stem cells collected and stored prior to receiving high-dose chemotherapy, the stem cells are then given back to the patient as a transplant. However, the use of high doses of chemotherapy is associated with significant side effects of nausea and vomiting. Before the use of newer medications, the incidence of nausea and vomiting could be as high as 70-90%.

Nausea is an unpleasant feeling and awareness of the urge to vomit. Vomiting is the process of throwing up forcefully the contents of the stomach. Retching is an act similar to vomiting but do not produce throwing up of the contents of the stomach. It is also called "dry heaves".

There are three kinds of nausea and vomiting associated with chemotherapy. Acute nausea and/or vomiting occur within the first 24 hours after administration of chemotherapy. Delayed nausea and/or vomiting begins after the first 24 hours of chemotherapy and could last for several days afterwards. Anticipatory nausea/vomiting is experienced prior to administration of the subsequent chemotherapy.

Chemotherapy produces nausea and vomiting by damaging the cells lining the stomach and intestines which results in the release a substance called serotonin. The serotonin binds to a protein or "receptor" (5-HT3 receptor) in the lining of the intestines. The receptors then send a message to the vomiting center in the brain. The brain then sends signals to the body to produce nausea and vomiting.

Another substance, called substance P, is also released from the lining of the stomach and intestines with damage by chemotherapy, and is released together with serotonin. The substance P binds to another protein called "neurokinin-1 receptor" or NK-1 receptor. These proteins are found in the intestines and another portion of the brain called "tractus solitarius". The brain then signals the body to produce nausea and vomiting.

The stimulation of the serotonin proteins results in acute nausea and vomiting. The stimulation of the NK-1 protein results in delayed nausea and vomiting.

There are medications that could block the serotonin and NK-1 proteins. Serotonin blockers such as ondansetron or Zofran® are now considered the medications of choice to prevent and treat nausea and vomiting in the transplant setting. However, their use could still result in nausea and vomiting in up to 40-50% of patients.

Nausea and vomiting negatively impacts the quality of life of patients undergoing stem cell transplant for their multiple myeloma and lymphoma. It can affect their appetite and sleep; and can interfere with activity, social life and enjoyment of life. Therefore, it is important to find better ways to prevent and control nausea and vomiting associated with chemotherapy.

There are two new medications that are available for patients who receive regular doses of chemotherapy. One is the long acting preparation of the serotonin blocker called palonosetron or Aloxi®. It is used to control both acute and delayed nausea and vomiting. Another medication could block the NK-1 receptor, and is called aprepitant or Emend®. This prevents delayed nausea and vomiting.

Although these two medications are tested and proven to be effective among patients who receive regular doses of chemotherapy, they have not been tested in combination among patients who undergo high doses of chemotherapy in the setting of autologous stem cell transplant.

The purpose of this study is to evaluate if the combination of these two medications, together with small doses of steroids (dexamethasone), would be effective in preventing both acute and delayed vomiting associated with high doses of chemotherapy and stem cell transplant for patients with multiple myeloma and lymphoma. The usual way to administer palonosetron is by single injection in the vein before chemotherapy. This is shown to be effective for chemotherapy given for 1 day. Since chemotherapy regimen for transplant requires multiple days of treatment, palonosetron will also be administered on multiple days thereby delivering higher doses of this drug. Aprepitant would be administered at standard doses. This study would assess if combining palonosetron and aprepitant as well as giving multiple and higher doses of palonosetron would be safe and effective in the control of nausea and vomiting in the setting of transplant. The study would evaluate the effect of combined palonosetron and aprepitant on the quality of life with regards to nausea and vomiting, of patients undergoing transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple myeloma and lymphoma deemed by the treating institution to be candidates for high dose chemotherapy and autologous hematopoietic stem cell transplant.
2. Both males and females are eligible.
3. Patients should be 18 years old; multiple myeloma patients up to age 75 and lymphoma patients up to age 65 are eligible.
4. Patients with Karnofsky performance status of 60% or better.
5. Patients should have at least 2.5 x 106 cyropreserved CD34+ cells per kilogram available for transplantation.
6. Patients with adequate bone marrow function as defined as ANC ≥1000 cells/mm3 , platelet ≥ 75,000 cells/mm3.
7. Lymphoma patient must have adequate renal function as defined by a calculated creatinine clearance of 50% measured in ml/min.
8. The criteria for renal function does not apply for multiple myeloma patients. Multiple myeloma patients undergoing hemodialysis are eligible.
9. All patients must have a MUGA scan indicating a left ventricular ejection fraction (LVEF) of greater or equal to 48% within 42 days prior to registration.
10. Patients must have adequate pulmonary function as defined by room air pulse oximetry equal to or greater than 93%, and pulmonary function tests (FEV1 and DLCO) equal to or greater than 50% of predicted values.
11. Patients with adequate hepatic function as defined by serum bilirubin lower than 2.5 mg/dL and liver function tests to not exceed greater than 1.5x of the institutions ULN.
12. All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with the institutional and federal guidelines.
13. Patients must be able to complete the anti-emesis assessment questionnaire. A Spanish questionnaire will be available for Hispanic-speaking patients.

Exclusion Criteria:

1. Patients with nausea and have emetic episodes, and are receiving any anti-emetic medication taken within 24 hours of receiving antibiotics.
2. Active infection involving intravenous antibiotics.
3. Patients with known active hepatitis B and/or hepatitis C infections are excluded.
4. Patients with known HIV infection.
5. Primary or secondary brain neoplasms with increased intracranial pressure.
6. Received intrathecal chemotherapy within 24 hours of first dose of conditioning chemotherapy.
7. Patients who are nursing mothers or pregnant. Females of childbearing age are required to have a negative serum B-HCG pregnancy test 24 hours prior to enrollment on the study.
8. Patients with previous malignancies at other sites except surgically treated nonmelanomatous skin cancers, prostate cancer or superficial cervical cancers, or other cancer from which the patient had been disease free for 5 or more years.
9. Patients with uncontrolled medical problems such as diabetes mellitus, cardiac (i.e. congestive heart failure, coronary heart disease, arrhythmias), pulmonary hepatic and renal disease unless renal insufficiency is felt to be secondary to multiple myeloma,
10. Myocardial infarction within 6 months of enrollment in the study.
11. Major surgery within 4 weeks of enrollment.
12. Morbid obesity (BMI>40)
13. Patients with psychiatric or central nervous systems disorders interfering with ability to comply with study protocol.
14. Patients receiving therapeutic anticoagulant therapy for venous thromboembolic episode or other hypercoaguable states. Coumadin at 1 mg as prophylaxis for central venous catheter is allowed.
15. Known hypersensitivity to 5-HT3 antagonists and Aprepitant and their components.
16. Use of non-prescription and herbal-type medications within 72 hours of enrollment on the study. Their use are not allowed during the study. Multivitamins, nutritional supplements such as Boost, and other electrolyte replacements are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Aljitawi, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients undergoing Autologous Stem Cell Transplant (ASCT) for multiple myeloma (MM) (n=10) and relapsed lymphoma (n=10) at the University of Kansas Medical Center were enrolled. 2 patients were excluded from analysis - both patients met exclusion criteria
Pre-assignment Details: Emetic responses were assessed by daily patient diaries and the Multinational Association for Supportive Care in Cancer Antiemetic Tool (MAT). Nausea was measured using a Nausea Visual Score (NVS) of 0 to 10 with score of 0 having no nausea. A "modified" Osoba module was used to assess quality of life (QOL).
Groups:
- Group A - Subjects With Multiple Myeloma: Group A: Subjects with Multiple Myeloma
  * Conditioning regimen, over a 7 day period, includes:
  * Melphalan 70-100 mg, Dexamethasone 4 mg IV push, Aprepitant 125 mg PO, Palonosetron 0.25 mg IV over 30 seconds, Aprepitant 80 mg PO, Dexamethasone 4 mg IV and Lorazepam 1 mg IV x 1 dose 30 minutes prior to stem cell infusion
- Group B - Subjects With Relpased Lymphoma: Group B: Subjects with Lymphoma
  * Conditioning regimen, over a 7 day period, includes: (BEAC)
  * carmustin (BCNU) 300 mg/m2 IV x 1,Cytarabine 100 mg/m2 IV BID, Etoposide 100 mg/m2 IV BID, administer after, Cyclophosphamide 35 mg/kg QD, Dexamethasone 4 mg IV push, Aprepitant 125 mg PO, Palonosetron 0.25 mg IV over 30 seconds, Aprepitant 80 mg PO, Lorazepam 1 mg IV x 1 dose 30 minutes prior to stem cell transplant
Period: Overall Study
Arm/Group | Group A - Subjects With Multiple Myeloma | Group B - Subjects With Relpased Lymphoma
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — history of malignancy within 5 years | 1 | 0
Not completed — History of prepartive regimen | 0 | 1

BASELINE CHARACTERISTICS:
Population: 2 patients excluded from analysis
Groups:
- Subjects With Multiple Myeloma: Group A: Subjects with Multiple Myeloma
  * Conditioning regimen, over a 7 day period, includes:
  * Melphalan 70-100 mg, Dexamethasone 4 mg IV push, Aprepitant 125 mg PO, Palonosetron 0.25 mg IV over 30 seconds, Aprepitant 80 mg PO, Dexamethasone 4 mg IV and Lorazepam 1 mg IV x 1 dose 30 minutes prior to stem cell infusion
  Group B: Subjects with Lymphoma
  * Conditioning regimen, over a 7 day period, includes: (BEAC)
  * BCNU 300 mg/m2 IV x 1,Cytarabine 100 mg/m2 IV BID, Etoposide 100 mg/m2 IV BID, administer after, Cyclophosphamide 35 mg/kg QD, Dexamethasone 4 mg IV push, Aprepitant 125 mg PO, Palonosetron 0.25 mg IV over 30 seconds, Aprepitant 80 mg PO, Lorazepam 1 mg IV x 1 dose 30 minutes prior to stem cell transplant
- Group B Lymphoma: Includes patients with Hodgkin's Disease and Non-Hodgkin's lymphoma
- Total: Total of all reporting groups
Arm/Group | Subjects With Multiple Myeloma | Group B Lymphoma | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
emetic response, adverse events, quality of care [Median (Full Range); unit: participants] | 9 [0 to 9] | 9 [0 to 9] | 9 [0 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Overall Emetic Response: Acute
Description: Complete Control (CC) - no emetic episode in 24 hours, no rescue medications and nausea visual scale (NVS) of ≤ 2.5, Complete Emetic Response (CR) - 0 emetic episodes, no rescue medications. Major Emetic Response (MR) - 0 to 2 emetic episodes within 24 hour period with or without rescue medications.
  Minor Emetic Response (mR) - 3 to 5 emetic episodes within 24 hour period with or without rescue medications.
  Failure - >5 emetic episodes within 24 hour period. No Significant Nausea (NSN) - maximum NVS ≤ 5.
Time Frame: 24 hours after chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Subjects With Multiple Myeloma | Group B - Subjects With Relpased Lymphoma
Number analyzed (Participants) | 9 | 9
Participants
  CC | 5 | 9
  CR | 1 | 0
  MR | 3 | 0
  mr | 0 | 0
  Failure | 0 | 0
  NSN | 9 | 9

2. Primary Outcome: Overall Emetic Response: Delayed
Description: as for outcome 1
Time Frame: 24 to 72 hours after chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Subjects With Multiple Myeloma | Group B - Subjects With Relpased Lymphoma
Number analyzed (Participants) | 9 | 9
Participants
  CC | 2 | 4
  CR | 1 | 0
  MR | 6 | 5
  mR | 0 | 0
  Failure | 0 | 0
  NSN | 0 | 8

3. Primary Outcome: Overall Emetic Response: Extended
Description: as for outcome 1
Time Frame: 72 hours after chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Subjects With Multiple Myeloma | Group B - Subjects With Relpased Lymphoma
Number analyzed (Participants) | 9 | 9
Participants
  CC | 1 | 2
  CR | 0 | 0
  MR | 7 | 7
  mR | 0 | 0
  Failure | 0 | 0
  NSN | 0 | 5

4. Primary Outcome: Overall Emetic Response
Description: Clinical responses were summarized using frequencies and percentages by phase, disease group, and overall. To compute emetic response by phase, the previously defined criteria were applied to each day of the three phases independently. The worst response was used to represent the response in each of these phases and overall emetic response. Overall emetic response was computed by applying the same definitions of emetic response to the entire study period.
Time Frame: At leaset 24 hours to more than 72 hours after chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Subjects With Multiple Myeloma | Group B - Subjects With Relpased Lymphoma
Number analyzed (Participants) | 9 | 9
Participants
  CC | 0 | 1
  CR | 0 | 0
  MR | 8 | 6
  mR | 1 | 2
  Failure | 0 | 0
  NSN | 6 | 5

5. Secondary Outcome: Impact of Nausea and Vomiting on the Quality of Life of Patients Undergoing Autologous HSCT
Description: To determine quality of life, subjects' responses to the modified Osoba modules were converted to a 0 - 100 scale, with higher scores indicative of better QOL
Time Frame: 24 hours, Day 3, Day 7
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day +30
Groups:
- Subjects With Multiple Myeloma: Group A: Subjects with Multiple Myeloma
  * Conditioning regimen, over a 7 day period, includes:
  * Melphalan 70-100 mg, Dexamethasone 4 mg IV push, Aprepitant 125 mg PO, Palonosetron 0.25 mg IV over 30 seconds, Aprepitant 80 mg PO, Dexamethasone 4 mg IV and Lorazepam 1 mg IV x 1 dose 30 minutes prior to stem cell infusion
- Patients With Lymphoma: Group B: Subjects with Lymphoma
  * Conditioning regimen, over a 7 day period, includes: (BEAC)
  * BCNU 300 mg/m2 IV x 1,Cytarabine 100 mg/m2 IV BID, Etoposide 100 mg/m2 IV BID, administer after, Cyclophosphamide 35 mg/kg QD, Dexamethasone 4 mg IV push, Aprepitant 125 mg PO, Palonosetron 0.25 mg IV over 30 seconds, Aprepitant 80 mg PO, Lorazepam 1 mg IV x 1 dose 30 minutes prior to stem cell transplant
Arm/Group | Subjects With Multiple Myeloma | Patients With Lymphoma
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/9 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Multiple Myeloma (N=9) | Patients With Lymphoma (N=9)
Infection, Abdomen NOS (Infections and infestations) | 0 (0) | 1 (1)
Gastric Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gallbladder pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Infection, Catheter-related (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No